CLINICAL TRIAL: NCT03699046
Title: Randomized Pilot Study Comparing the Effectiveness of Subchondroplasty Combined With Arthroscopy to Arthroscopy Alone for Treating Bone Marrow Lesions of the Knee
Brief Title: Evaluating the Effectiveness of Subchondroplasty for Treating Bone Marrow Lesions of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: McCaig Institute for Bone and Joint Health - Centre for Mobility and Joint Health (Unknown)
Responsible Party: Principal Investigator, Alexander Rezansoff, Orthopaedic Surgeon and Clinical Lecturer, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB18-0650
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee; Arthroscopy; Musculoskeletal Disease; Bone Marrow Edema; Subchondral Bone Edema; Knee Osteoarthritis
Keywords: Bone Marrow Lesion; Subchondroplasty; Knee Function; Knee Pain; Bone Quality; Bone Micro-architecture
MeSH Terms: conditions — Osteoarthritis, Knee; Musculoskeletal Diseases | interventions — Urocortins

STUDY DESIGN:
Intervention Model Description: The control group will be patients receiving knee arthroscopy alone and the intervention group will be patients receiving subchondroplasty and knee arthroscopy.
Who Masked: Participant
Masking Description: Patients will be randomized at the time of surgery to either the control group or the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Subchondroplasty and Knee Arthroscopy (Active Comparator): Patients randomized to the Subchondroplasty and Knee Arthroscopy group will receive the subchondroplasty procedure before or after knee arthroscopy that will be completed based on current standard of care guidelines.
  Interventions: Procedure: Subchondroplasty and Knee Arthroscopy; Biological: Subchondroplasty
- Knee Arthroscopy Alone (Sham Comparator): Patients randomized to the Knee Arthroscopy Alone group will receive the knee arthroscopy that will be completed based on current standard of care guidelines.
  Interventions: Procedure: Knee Arthroscopy Alone

INTERVENTIONS:
Procedure: Subchondroplasty and Knee Arthroscopy — Subchondroplasty® (SCP®) is a procedure performed along with minimally-invasive arthroscopy. The bone marrow lesion(s) will be located using pre-operative MRI combined with fluoroscopy (intra-operative X-ray) and a small, drillable AccuPort® Delivery Cannula will be placed in the appropriate position. The cannula will then be drilled into the bone marrow lesion(s) and a flowable, synthetic, calcium phosphate bone substitute (AccuFill® Bone Substitute Material, Zimmer Biomet) will be injected into the lesion(s). The calcium phosphate bone substitute will then harden, improve the structural integrity of the damaged subchondral bone, and will gradually be resorbed and replaced with new bone.
  Arms: Subchondroplasty and Knee Arthroscopy
Procedure: Knee Arthroscopy Alone — Knee arthroscopy is a surgical procedure that involves the orthopaedic surgeon making small incisions in the knee and then inserting a small camera into the joint. Following the insertion of the camera, multiple procedures can be completed to treat a number of different conditions such as repair or partial/complete removal of the meniscus, debridement, lavage, removal of a loose body among others.
  Arms: Knee Arthroscopy Alone
Biological: Subchondroplasty — Subchondroplasty® (SCP®) is a procedure performed along with minimally-invasive arthroscopy. The specific biological component of the procedure involves the injection of the AccuFill® Bone Substitute Material (Zimmer Biomet), which is a a flowable, synthetic, calcium phosphate bone substitute, into the bone marrow lesion(s).
  Other Names: SCP® (Zimmer)
  Arms: Subchondroplasty and Knee Arthroscopy

SUMMARY:
The primary objective of this randomized pilot study is to evaluate whether subchondroplasty combined with knee arthroscopy is more effective at reducing knee pain and improving knee function compared to knee arthroscopy alone. All knee function outcomes will be assessed at initial presentation, 3 months, 6 months, 12 months, and 24 months following surgery using validated questionnaires. Patient-reported pain will also be recorded at 2 weeks after surgery.

The secondary objective of the study is to determine whether the subchondroplasty and knee arthroscopy group has better bone quality and bone micro-architecture compared to the group receiving knee arthroscopy alone. Bone quality/micro-architecture will be evaluated at baseline, 3 months, and 12 months following surgery using Magnetic resonance imaging (MRI) and High-Resolution Peripheral Quantitative CT (HR-pQCT) imaging and at baseline, 3 months, 12 months, and 24 months after surgery using X-rays.

DETAILED DESCRIPTION:
The investigators hypothesize that patients receiving subchondroplasty combined with arthroscopy will have reduced knee pain, improved knee function, and improved bone quality and micro-architecture compared to patients receiving arthroscopy alone who have symptomatic early osteoarthritis with the presence of at least one BML observed on MRI.

Patients who provide informed consent to enroll in the study will be scheduled for knee surgery and randomized to receive subchondroplasty and arthroscopy or arthroscopy alone. Knee function outcomes will be assessed at initial presentation, 3 months, 6 months, 12 months, and 24 months following surgical intervention. Patient-reported pain will also be recorded at 2 weeks following surgical intervention. The evaluation of bone quality and micro-architecture will occur at baseline, 3 months, and 12 months following surgical intervention. X-rays will also be evaluated at the 24-month time-point.

ELIGIBILITY:
Inclusion Criteria:

1. 40 years of age or older
2. Kellgren-Lawrence grade 1-3 osteoarthritis in the affected knee
3. Has experienced pain in the affected knee for at least 3 months
4. Candidate for knee arthroscopy (moderate to severe symptoms, lack of response to non-operative care, and/or mechanical symptoms)
5. Stable ligament exam
6. No additional injuries affecting the study knee or contralateral knee
7. Candidate for MRI (no pacemaker, aneurysmal clip, eye prosthesis, pregnancy, neurostimulator, implanted stimulator [e.g. diabetes pump])
8. Confirmed visualization of at least 1 bone marrow lesions using T2 weighted MRI

Exclusion Criteria:

1. Determined to not be a surgical candidate
2. Kellgren-Lawrence grade 4 osteoarthritis
3. Unable to fit in XtremeCT scanner (based on measurement at time of recruitment)
4. Contraindications to MRI
5. Any hardware present in either knee that could interfere with MRI signal
6. Bone marrow lesion(s) caused by acute trauma prior to enrolment
7. Radiographic mal-alignment defined by obvious valgus > 7° or obvious varus > 7° on measured hip-knee-ankle angle
8. No bone marrow lesion detected on baseline (pre-operative) MRI
9. Rheumatoid arthritis
10. Septic arthritis
11. Reactive arthritis
12. Gout
13. Osteochondritis dissecans of knee resulting in significant bone loss
14. Collapse of subchondral bone
15. Restricted knee range of motion: passive flexion < 110° or a flexion contracture > 30°
16. Ligament instability in either knee
17. History of other arthropathies (e.g. sickle cell or autoimmune disease)
18. History of uncontrolled diabetes: HbA1C level of 8 or higher, measured within 3 months of enrollment
19. Unable to perform a functional assessment of either knee
20. Current smoker or stopped smoking for less than 3 months
21. History of invasive malignancy (Unless treated in the past and has had no clinical signs or symptoms of malignancy for 5 years or longer)
22. Has a primary bone tumor in the knee or adjacent to the knee
23. Having surgery on another part of the lower limb in addition to the study procedure
24. Taking prescription pain medication other than NSAIDs or acetominophen
25. Active infection or a history of joint infection
26. Pursuing action through the Workers' Compensation Board - Alberta
27. BMI > 40

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire scores | Baseline (pre-surgery), 3 months, 6 months, 12 months, 24 months post-surgery.
  The primary outcome measure will be the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire scores for knee pain and knee function.
  The KOOS questionnaire consists of 5 different sub-scales including Symptoms (7 questions), Pain (9 questions), Activities of Daily Living (17 questions), Sports/Recreation (5 questions), and Quality of Life (4 questions). A normalized score from 0-100 (100 indicates no problems/symptoms and 0 indicates extreme problems/symptoms) is calculated for each sub-scale individually.

SECONDARY OUTCOMES:
Change in International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form scores | Baseline (pre-surgery), 3 months, 6 months, 12 months, 24 months post-surgery.
  Knee pain and function will also be evaluated using the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form scores.
  The IKDC includes three different domains including Symptoms (7 questions), Sports Activities (2 questions, 1 multi-part question), and Function (1 multi-part question). A total score from 0-100 (100 indicates no problems/symptoms and 0 indicates extreme problems/symptoms) is calculated.
Change in Patient-Reported Pain scores on the Visual Analog Scale (VAS) | Baseline (pre-surgery), 2 weeks, 3 months, 6 months, 12 months, 24 months post-surgery.
  Knee pain will also be evaluated using the Visual Analog Scale (VAS) scores for patient-reported pain.
  The Visual Analog Scale (VAS) consists of a 10 cm long straight line that starts from the lowest value of 0 (no pain) at one end, and the highest value of 10 (worst pain possible) at the other. Patients are asked to mark a place on the line that represents the severity of their pain. Scores are recorded in millimetres from 0-100 with 0 indicating no pain and 100 indicating the worst pain possible.
Change in bone quality/micro-architecture evaluated using magnetic resonance imaging (MRI) | Baseline (pre-surgery), 3 months, 12 months post-surgery
  The bone quality and micro-architecture of the bone marrow lesion(s) in the knee, and the knee overall, will be evaluated using magnetic resonance imaging (MRI). MRI will be used to identify the presence of bone marrow lesion(s) in the knee at baseline before surgery using a T2 weighted fat-suppression sequence and evaluate the bone marrow lesion(s) post-surgery.
Change in bone quality/micro-architecture evaluated using High-Resolution Peripheral Quantitative CT (HR-pQCT) imaging | Baseline (pre-surgery), 3 months, 12 months post-surgery
  The bone quality and micro-architecture of the bone marrow lesion(s) in the knee, and the knee overall, will also be evaluated using High-Resolution Peripheral Quantitative CT (HR-pQCT) imaging. HR-pQCT imaging will be used to evaluate the bone micro-architecture of the knee and the bone marrow lesion(s) before and after surgery.
Change in bone quality/micro-architecture evaluated using X-rays | Baseline (pre-surgery), 3 months, 12 months, 24 months post-surgery.
  The bone quality and micro-architecture of the bone marrow lesion(s) in the knee, and the knee overall, will also be evaluated using X-ray. X-ray imaging will be used to evaluate bone quality and osteoarthritis status before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rezansoff, MD, FRCSC, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada